CLINICAL TRIAL: NCT02592863
Title: A Double-Blind, Placebo-Controlled, Randomized Trial of Pentoxifylline for Imbalance Secondary to Insufficient Microvascular Perfusion
Brief Title: Trental for the Treatment of Vertigo/Dizziness/Imbalance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Placebo effect
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Arnaldo L. Rivera, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1214160
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dizziness; Vertigo
MeSH Terms: conditions — Dizziness; Vertigo | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pentoxifylline (Experimental): Patients will take Trental (Pentoxifylline) 3 times per day for 12 weeks
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Patients will take placebo 3 times per day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Patients will take Trental (Pentoxifylline) 3 times per day for 12 weeks
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — Patients will take placebo 3 times per day for 12 weeks
  Arms: Placebo

SUMMARY:
Imbalance, dizziness and vertigo as a result of problems in the inner ear (vestibular dysfunction) are becoming increasingly more prevalent in Americans 40 years of age and older. The symptoms have a severe impact on affected individuals with detrimental effects on work, travel, social and family life. These patients see doctors often with no relief in their symptoms.

The most promising help for these patients is to use medication that will increase blood flow to the inner ear. Pentoxifylline (Trental) has been shown to increase microvascular blood flow.

DETAILED DESCRIPTION:
One potential cause of vestibular dysfunction is a decrease in or insufficient blood flow to the inner ear. Studies have shown that when the blood flow is decreased to the inner ear, patients will become dizzy and off balance. This study will use validated instruments to evaluate the effectiveness of Trental in patients that present to our providers with vertigo, dizziness, or imbalance and meet inclusion criteria. They will be blinded and randomized to treatment or placebo, which they will take for ~12 weeks. Patients will completed validated surveys 3 times (beginning, middle and end of study) as well as account for the number of times they have fallen and if they have missed any work due to their symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 40 years and older
2. English as primary language
3. Diagnosis of multisensory losses, presbystasis, bilateral vestibulopathy, central vascular insufficiency, small vessel circulatory disease, generalized imbalance, and idiopathic peripheral vertigo scoring at least 16 on the Dizziness Handicap Inventory
4. Willingness to complete surveys and take medication as prescribed

Exclusion Criteria:

1. Diagnosis of the following: benign paroxysmal positional vertigo, Meniere's disease, vestibular migraine with headache, intracranial mass, perilymphatic fistula, or multiple sclerosis
2. history of cholesteatoma
3. Prior ear surgery other than myringotomy and tube placement
4. Prior radiation to head or neck
5. previous use of vestibulotoxic medications where the enrolling provider determines the drug exposure to be the cause of imbalance
6. Use of blood thinning medications
7. intolerance/allergy to pentoxifylline or methylxanthines, as well as recent cerebral or retinal hemorrhage (past 3 months)
8. Pregnant or lactating females.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo E Rivera, M.D., Principal Investigator — University of Missouri - Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 10 | 16
Completed | 7 | 13
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: We only evaluated patients that completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 6 | 10 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 3 | 8 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 12 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Effect of Trental Treatment Using the Dizziness Handicap Inventory, Vestibular Activities and Participation, and European Evaluation of Vertigo Scale
Description: The Dizziness Handicap Inventory (DHI) is 25 question self report questionnaire that measures how dizziness affects a person's daily life. The questions are grouped into three domains: physical (P), emotional (E), and functional (F). Each question has three possible answers: "Always", "Sometimes", or "No". The answers are worth points, with "Always" being worth 4 points, "Sometimes" worth 2 points, and "No" worth 0 points. After answering all the questions, the total score is calculated, ranging from 0 to 100 points. A higher score indicates a more severe handicap, with 0 points indicating no effect and 100 points indicating maximum effect.
Time Frame: 12 weeks
Population: Determine the effect of 12 weeks of Trental compared to Placebo in patients with reported dizziness on the Dizziness Handicap Inventory
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 7 | 13
Score on a scale
  Baseline DHI | 46.57 (16.236) | 53.85 (22.825)
  End of Treatment DHI | 36.57 (20.582) | 42.83 (22.262)

2. Primary Outcome: Effect of Trental Treatment Using the European Evaluation of Vertigo Scale
Description: The European Evaluation of Vertigo scale (EEV) is a physician-administered questionnaire that only assesses symptoms of the vestibular syndrome: illusion of movement, duration of illusion, motion intolerance, neurovegetative signs, and instability. The symptoms are ranked on a scale of 0 (no problem) to 4 (severe problem) and each area of assessment is stand alone (meaning the scores from each area to do not combine to create one larger score)
Time Frame: 12 Weeks
Population: Determine the effect of 12 weeks of Trental compared to Placebo in patients with reported dizziness on the European Evaluation of Vertigo scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 7 | 13
units on a scale
  Baseline EEV - Illusion of Movement | 2.00 (1.155) | 2.62 (0.768)
  End of Treatment (EOT) - Illusion of movement | 1.57 (1.272) | 1.55 (1.128)
  Baseline EEV - Duration of Illusion | 2.00 (1.291) | 2.46 (1.127)
  EOT EEV - Duration of Illusion | 1.43 (0.787) | 1.64 (1.206)
  Baseline EEV - Motion Intolerance | 0.86 (1.464) | 0.69 (0.947)
  End of Treatment EEV - Motion Intolerance | 0.57 (1.134) | 0.55 (0.934)
  Baseline EEV - Neurovegetative | 0.14 (0.378) | 0.92 (1.256)
  End of Treatment EEV - Neurovegetative | 0 (0) | 0.45 (1.036)
  Baseline EEV - Instability | 2.29 (0.756) | 2.46 (0.776)
  EOT - Instability | 1.0 (0.816) | 1.145 (0.820)

3. Primary Outcome: Effect of Trental Treatment Using the Vestibular Activities and Participation Survey
Description: Vestibular Activities and Participation (VAP) is 34-item self-report tool that measures the extent of activity limitations and participation restrictions caused by vestibular disorders. The VAP can be used for assessment, intervention planning, outcome evaluation, and to reflect a patient's status. Answers are ranked on a likert scale where 0 is no problem and 4 is unable to do. Scores are averaged and the higher the score the worse the problem, such that 0 is no problem and 54 or great is a severe problem.
Time Frame: 12 Weeks
Population: Determine the effect of 12 weeks of Trental compared to Placebo in patients with reported dizziness on Vestibular Activities and participation survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 7 | 13
score on a scale
  Baseline VAP | 1.487 (0.5914) | 1.405 (0.5894)
  End of treatment VAP | 1.12 (0.642) | 1.02 (0.809)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Definition of adverse event and/or serious adverse event is not different than that published on clinicaltrials.gov.
Arm/Group | Pentoxifylline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 0/7 | 0/13

LIMITATIONS AND CAVEATS:
Early termination due to placebo effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT02592863/Prot_SAP_000.pdf